CLINICAL TRIAL: NCT05309837
Title: A Two-center, Randomized, Double-blind, Placebo Controlled, Parallel Study to Evaluate the Effect of Polydextrose on Fecal Bulk and Bowel Function in Mildly Constipated Subjects
Brief Title: Effect of Polydextrose on Fecal Bulk and Bowel Function in Mildly Constipated Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tate & Lyle (Industry)
Collaborators: Oy Foodfiles Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TALI "4010"
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Constipation; Gastrointestinal Dysfunction
Keywords: polydextrose; mild constipation; faecal bulk; bowel function; clinical trial; fibre
MeSH Terms: conditions — Constipation | interventions — polydextrose

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polydextrose (PDX) (Active Comparator): Subject consumed a daily dose of 18g polydextrose enriched drink mixtures and biscuits (12 g from the drink mixtures and 6 g from the biscuits) providing 16.2 g dietary fibre/d.
  Interventions: Dietary Supplement: Polydextrose
- Control (CON) (Placebo Comparator): Subjects consumed placebo products, where maltodextrin replaced PDX and differed only in the amount of fibre per gram (1.7 g).
  Interventions: Dietary Supplement: placebo-controlled

INTERVENTIONS:
Dietary Supplement: Polydextrose — Polydextrose-enriched food products
  Arms: Polydextrose (PDX)
Dietary Supplement: placebo-controlled — Control food products
  Arms: Control (CON)

SUMMARY:
Polydextrose (PDX) (8-30g/day) has been reported to increase faecal bulk and consistency, leading to easier stool passage in healthy subjects. Studies on its effect on defaecation frequency and colonic transit time have provided mixed results. The primary objective was to investigate the effect of PDX consumption by mildly constipated subjects on faecal bulk, measured as total faecal wet weight of 4-day collections. Secondary outcomes (faecal dry weight, defaecation frequency, stool consistency, ease of stool passage, total colonic transit time and gastrointestinal symptoms) were also explored. 51 subjects participated in a 4-week, two-center, randomized, double-blind, placebo-controlled, parallel study testing a control (CON) and a PDX treatment (18 g/d included in biscuits and drink mixtures)

ELIGIBILITY:
Inclusion Criteria:

1. Mildly constipated healthy adults (who defecate 3- 5 days per week assessed by a 7-day bowel diary)
2. Provision of signed and dated informed consent prior to any study procedures
3. Body mass index (BMI) ≥ 19 and ≤ 29 kg/m2 at the screening visit
4. Total score on fibre intake questionnaire max 17 points for women and 20 points for men (where each point represents approximately 1 g fibre intake)
5. Use of adequate contraception in females of childbearing potential

Exclusion Criteria:

1. Regular use of laxatives
2. Use of medication which alters study subjects' gastrointestinal function (e.g. including but not exclusive neuroleptic medication, medication for Parkinson disease, opioids)
3. History of digestive disease (e.g. celiac disease, Crohn's disease, ulcerative colitis, gastrointestinal malignancy, fistula of intestine, ischemic colitis, bile acid malabsorption, repeated diverticulitis)
4. Type I and II diabetes
5. Previous major gastrointestinal surgery (e.g. intestinal resection, total gastrectomy, subtotal gastrectomy) or surgical treatment of obesity (within 6 months before the screening visit)
6. Present cancer (except basal cell skin cancer or squamous cell skin cancer, carcinoma in situ)
7. Untreated thyroid disease
8. History of stroke or myocardial infarction within six months prior the screening visit
9. Subjects who were actively dieting for weight loss, or had eating disorders (anorexia, bulimia)
10. Lack of compliance to the study procedures
11. Females who were pregnant or breast-feeding or planning pregnancy
12. Known or suspected abuse of alcohol (more than 14 units of alcohol per week, one unit = 4 cl spirit, 12 cl wine or 33 cl medium strong beer / cider),
13. Allergy/hypersensitivity/intolerance to study products
14. Vegetarians or regularly consuming fibre supplements/fibre supplemented foods
15. Any clinically significant disease/condition which in the Investigator's opinion could interfere with the results of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-09-19 (Actual)

PRIMARY OUTCOMES:
Faecal bulk | 4-day collections
  Measured as total faecal wet weight

SECONDARY OUTCOMES:
Faecal dry weight | 4-day collections during the intervention period
  Measured as total faecal dry weight
Defaecation frequency | 7-day period during the run-in period and intervention period
  Recorded as defaecation frequency (i.e. number of stools)
Stool consistency | 7-day period during the run-in period and intervention period
  Measured using the Bristol Stool Form (BSF) score (1 = separate hard lumps, like nuts (difficult defaecation), 2 = sausage shaped but lumpy, 3 = like a sausage or snake but with cracks on its surface, 4 = like a sausage or snake, smooth and soft, 5 = soft blobs with clear cut edge, 6 = fluffy pieces with ragged edges, a mushy stool, 7 = watery, no solid pieces)
Ease of stool passage | At the end of the intervention period
  Using a five-point scale (1 = very easy, 2 = easy, 3 = neither easy nor difficult, 4 = difficult, 5 = very difficult)
Total colonic transit time | At the end of the intervention period for three consecutive days
  Using radio-opaque, barium sulfate impregnated polyethylene pellets located inside gelatin capsules
Gastrointestinal symptoms | Once at the end of the intervention period and during the previous one week (7 day-period).
  Subjects ranked ranked the subjective tolerance variables daily to burping, cramping, distension/bloating, flatulence, nausea, reflux (heartburn) and vomiting on a four-point scale (1 = none, 2 = mild, 3 = moderate, 4 = severe)

CONTACTS AND LOCATIONS:
Overall Officials: Essi Sarkkinen, PhD, Study Director — Oy Foodfiles Ltd

IPD SHARING:
Plan to Share IPD: No